CLINICAL TRIAL: NCT00783432
Title: Active-Controlled Trial of the Safety and Tolerability of a MP03-33 in Patients With Chronic Allergic or Nonallergic Rhinitis
Brief Title: Study to Evaluate the Safety and Tolerability of a Nasal Spray in Patients With Chronic Allergic or Nonallergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Harry Sacks, MD, Vice President, Medical and Scientific Affairs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP432
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2009-10-02 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Allergic Rhinitis; Nonallergic Rhinitis
MeSH Terms: interventions — azelastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Astepro Nasal Spray (0.1% azelastine hydrochloride)
  Interventions: Drug: Astepro Nasal Spray (0.1% azelastine hydrochloride)
- 2 (Active Comparator): Astelin Nasal Spray (0.1% azelastine hydrochloride)
  Interventions: Drug: Astelin Nasal Spray (0.1% azelastine hydrochloride)

INTERVENTIONS:
Drug: Astepro Nasal Spray (0.1% azelastine hydrochloride) — 548 mcg (2 sprays per nostril) twice a day
  Arms: 1
Drug: Astelin Nasal Spray (0.1% azelastine hydrochloride) — 548 mcg (2 sprays per nostril) twice a day
  Arms: 2

SUMMARY:
The purpose of this study is to determine if Astepro Nasal Spray (0.1% azelastine hydrochloride) is as safe as Astelin Nasal Spray (0.1% azelastine hydrochloride)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 12 years of age and older with an established history (> 1 year) of rhinitis due to perennial allergies, non-allergic triggers or vasomotor rhinitis (VMR).
2. Provide written informed consent/pediatric assent. If the patient is a minor, a parent or legal guardian must give written informed consent
3. Willing and able to comply with the study requirements, including daily use of medication for a one year period, even if symptoms are not bothersome.
4. General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer
5. Patients receiving immunotherapy (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimen following a brief period of missed injections does not preclude participation)

Exclusion Criteria:

1. The use of any investigational drug within 30 days prior to screening. No other investigational products are permitted for use during the conduct of this study
2. Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose (Splenda® brand sweetener)
3. Women who are pregnant or nursing
4. Women of childbearing potential who are not abstinent and not practicing a medically acceptable method of contraception. Female patients must practice an acceptable contraceptive technique for 30 days before randomization and agree to continue its use during treatment and for 30 days after the last dose of study drug. Oral, intrauterine, implantable, injectable contraceptives, or a double barrier form of contraception are acceptable and the medication including dose, device or method must have been stable for at least 30 days before the first dose of study drug.
5. Nasal disease(s) likely to affect deposition of intranasal medication, such as sinusitis,rhinitis medicamentosa or clinically significant nasal polyposis or nasal structural abnormalities
6. Patients with asthma (with the exception of mild, intermittent asthma) or other significant pulmonary disease such as Chronic Obstructive Pulmonary Disease
7. Patients with a known history of alcohol or drug abuse
8. Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor, might significantly alter the evaluation of study
9. Clinically relevant abnormal history and/or physical findings which, in the opinion of the investigator or sponsor, would interfere with the objectives of the study or that may preclude compliance with the study procedures
10. Study site staff, immediate relatives of study site staff, or other individuals who would have access to the clinical study protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M. Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (1):
- Meda Clinical Trials Contact Center, Somerset, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First observation 24 July 2006 and last observation 28 Dec 2007
Pre-assignment Details: Subjects participated in a one-week screening period to identify appropriate subjects based on symptom scores
Groups:
- Astepro Nasal Spray; Astelin Nasal Spray: (0.1% azelastine hydrochloride)
Period: Overall Study
Arm/Group | Astepro Nasal Spray | Astelin Nasal Spray
Started | 430 (This includes 2 subjects that received a randomization number but did not receive study drug) | 432 (This includes 2 subjects that received a randomization number but did not receive study drug)
Completed | 345 | 354
Not Completed | 85 | 78
Not completed — Adverse Event | 22 | 17
Not completed — Lack of Efficacy | 20 | 21
Not completed — Lost to Follow-up | 11 | 6
Not completed — Withdrawal by Subject | 23 | 20
Not completed — subject moved | 3 | 5
Not completed — Protocol Violation | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Astepro Nasal Spray | Astelin Nasal Spray | Total
Number analyzed (Participants) | 428 | 430 | 858
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 10 | 21
  Between 18 and 65 years | 389 | 391 | 780
  >=65 years | 28 | 29 | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 41.2 (14.95) | 41.3 (15.12) | 41.2 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 236 | 457
  Male | 207 | 194 | 401
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 16 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 4 | 10
  White | 410 | 405 | 815
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Australia | 40 | 39 | 79
  Europe | 388 | 391 | 779
Duration of Rhinitis [Mean (Standard Deviation); unit: years] | 10.5 (11.04) | 11.3 (10.85) | 10.9 (10.95)
Total Nasal Symptom Score (AM + PM) [Mean (Standard Deviation); unit: units on a scale (0-3)] — TNSS scale: 0=no symptoms, 1=mild symptoms, 2=moderate symptoms and 3 = severe symptoms scored twice daily such that the maximum daily score is 24.
  units on a scale (0-3) | 9.69 (4.506) | 9.96 (4.725) | 9.82 (4.617)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events
Description: An AE can be any unfavorable and unintended sign,symptom, or disease temporally associated with the use of this investigational product, whether or not considered related to the investigational product. An AE is any untoward medical occurrence in a subject which does not necessarily have a causal relationship with this treatment.
Time Frame: 12 months
Population: Number of participants for analysis was based on a safety population that included any subject who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Astepro Nasal Spray | Astelin Nasal Spray
Number analyzed (Participants) | 428 | 430
Participants | 207 | 211

2. Primary Outcome: Focused Examination of the Head and Neck With Findings Recorded on a Numeric Scale.
Description: Examination of head and neck(scale: 0, 1+=Mild, 2+=Moderate, 3++Severe) for mucosal edema, nasal discharge, mucosal erythema, mucosal bleeding, mucosal ulcerations, crusting of mucosa, conjunctiva, tympanic membranes, lymph nodes of head and neck. Direct visual nasal examination (scale: None, Grade 2, Grade 3, and Grade 4) for epistaxis,ulceration and pain.
Time Frame: baseline and 12 months/ET
Measure: Number; unit: Participants
Arm/Group | Astepro Nasal Spray | Astelin Nasal Spray
Number analyzed (Participants) | 428 | 430
Participants
  Conjunctiva: Total baseline | 428 | 430
  Conjunctiva: baseline-None | 264 | 254
  Conjunctiva: baseline-Mild (1+) | 99 | 109
  Conjunctiva: baseline-Moderate (2+) | 53 | 54
  Conjunctiva: baseline-Severe (3+) | 12 | 13
  Conjunctiva: Total M12/ET | 414 | 417
  Conjunctiva: M12/ET-None | 366 | 363
  Conjunctiva: M12/ET-Mild (1+) | 44 | 43
  Conjunctiva: M12/ET-Moderate (2+) | 4 | 11
  Conjunctiva:M12/ET-Severe (3+) | 0 | 0
  Tympanic membranes: Total baseline | 428 | 430
  Tympanic membranes: baseline-None | 342 | 344
  Tympanic membranes: baseline-Mild (1+) | 60 | 62
  Tympanic membranes:baselineModerate (2+) | 21 | 17
  Tympanic membranes: baseline-Severe (3+) | 5 | 7
  Tympanic membranes: Total M12/ET | 414 | 417
  Tympanic membranes: M12/ET-None | 405 | 408
  Tympanic membranes:M12/ET-Mild (1+) | 8 | 5
  Tympanic membranes: M12/ET-Moderate (2+) | 1 | 4
  Tympanic membranes:M12/ET Severe (3+) | 0 | 0
  Lymphadenopathy: Total baseline | 428 | 430
  Lymphadenopathy: baseline-None | 389 | 393
  Lymphadenopathy: baseline-Mild (1+) | 32 | 27
  Lymphadenopathy: baseline-Moderate (2+) | 7 | 7
  Lymphadenopathy: baseline-Severe (3+) | 0 | 3
  Lymphadenopathy: Total M12/ET | 414 | 417
  Lymphadenopathy: M12/ET-None | 408 | 407
  Lymphadenopathy:M12/ET-Mild (1+) | 6 | 10
  Lymphadenopathy:M12/ET-Moderate (2+) | 0 | 0
  Lymphadenopathy: M12/ET-Severe (3+) | 0 | 0
  Mucosal edema: Total baseline | 428 | 430
  Mucosal edema: baseline-None | 32 | 30
  Mucosal edema: baseline-Mild (1+) | 91 | 80
  Mucosal edema: baseline-Moderate (2+) | 191 | 200
  Mucosal edema: baseline-Severe (3+) | 114 | 120
  Mucosal edema: Total M12/ET | 414 | 417
  Mucosal edema:M12/ET-None | 160 | 147
  Mucosal edema: M12/ET-Mild (1+) | 176 | 182
  Mucosal edema: M12/ET-Moderate (2+) | 69 | 76
  Mucosal edema: M12/ET-Severe (3+) | 9 | 12
  Nasal discharge: Total baseline | 428 | 430
  Nasal discharge: baseline-None | 40 | 44
  Nasal discharge: baseline-Mild (1+) | 113 | 109
  Nasal discharge: baseline-Moderate (2+) | 179 | 183
  Nasal discharge: baseline-Severe (3+) | 96 | 94
  Nasal discharge: Total M12/ET | 414 | 417
  Nasal discharge:M12/ET-None | 178 | 173
  Nasal discharge: M12/ET-Mild (1+) | 188 | 183
  Nasal discharge: M12/ET-Moderate (2+) | 46 | 54
  Nasal discharge:M12/ET-Severe (3+) | 2 | 7
  Mucosal erythema: Total baseline | 428 | 430
  Mucosal erythema: baseline-None | 80 | 82
  Mucosal erythema: baseline-Mild (1+) | 120 | 112
  Mucosal erythema: baseline-Monderate (2+) | 171 | 178
  Mucosal erythema: baseline-Severe (3+) | 57 | 58
  Mucosal erythema: Total M12/ET | 414 | 417
  Mucosal erythema: M12/ET-None | 213 | 221
  Mucosal erythema: M12/ET-Mild (1+) | 152 | 153
  Mucosal erythema: M12/ET-Moderate (2+) | 45 | 35
  Mucosal erythema:M12/ET-Severe (3+) | 4 | 8
  Mucosal bleeding: Total baseline | 428 | 430
  Mucosal bleeding: baseline-None | 362 | 376
  Mucosal bleeding: baseline-Mild (1+) | 56 | 51
  Mucosal bleeding: baseline-Moderate (2+) | 10 | 2
  Mucosal bleeding: baseline-Severe (3+) | 0 | 1
  Mucosal bleeding: Total M12/ET | 414 | 417
  Mucosal bleeding: M12/ET-None | 402 | 403
  Mucosal bleeding: M12/ET-Mild (1+) | 11 | 10
  Mucosal bleeding: M12/ET-Moderate (2+) | 1 | 4
  Mucosal bleeding: M12/ET-Severe (3+) | 0 | 0
  Mucosal ulcerations: Total baseline | 428 | 430
  Mucosal ulcerations: baseline-None | 348 | 362
  Mucosal ulcerations: baseline-Mild (1+) | 48 | 37
  Mucosal ulcerations: baseline-Moderate (2+) | 26 | 25
  Mucosal ulcerations: baseline-Severe (3+) | 6 | 6
  Mucosal ulcerations: Total M12/ET | 414 | 417
  Mucosal ulcerations: M12/ET-None | 401 | 404
  Mucosal ulcerations: M12/ET-Mild (1+) | 11 | 10
  Mucosal ulcerations: M12/ET-Moderate (2+) | 2 | 3
  Mucosal ulcerations: M12/ET-Severe (3+) | 0 | 0
  Crusting of mucosa: Total baseline | 428 | 430
  Crusting of mucosa: baseline-None | 293 | 311
  Crusting of mucosa: baseline-Mild (1+) | 86 | 75
  Crusting of mucosa: baseline-Moderate (2+) | 36 | 35
  Crusting of mucosa: baseline-Severe (3+) | 13 | 9
  Crusting of mucosa: Total M12/ET | 414 | 417
  Crusting of mucosa: M12/ET-None | 387 | 382
  Crusting of mucosa: M12/ET-Mild (1+) | 24 | 32
  Crusting of mucosa: M12/ET-Moderate (2+) | 3 | 3
  Crusting of mucosa:M12/ET-Severe (3+) | 0 | 0
  Epistaxis: Total baseline | 428 | 430
  Epistaxis: baseline None | 402 | 416
  Epistaxis: baseline Grade 2 | 26 | 12
  Epistaxis: baseline Grade 3 | 0 | 1
  Epistaxis: baseline Grade 4 | 0 | 1
  Epistaxis:Total M12/ET | 414 | 417
  Epistaxis: M12/ET None | 413 | 415
  Epistaxis: M12/ETGrade 2 | 1 | 2
  Epistaxis:M12/ET Grade 3 | 0 | 0
  Epistaxis: M12/ETGrade 4 | 0 | 0
  Ulceration: Total baseline | 428 | 430
  Ulceration: baseline None | 365 | 373
  Ulceration: baseline Grade 2 | 63 | 57
  Ulceration: baseline Grade 3 | 0 | 0
  Ulceration: baseline Grade 4 | 0 | 0
  Ulceration: Total M12/ET | 413 | 417
  Ulceration:M12/ET None | 404 | 411
  Ulceration: M12/ET Grade 2 | 8 | 6
  Ulceration: M12/ET Grade 3 | 1 | 0
  Ulceration: M12/ET Grade 4 | 0 | 0
  Pain: Total baseline | 428 | 430
  Pain: baseline None | 377 | 382
  Pain: baseline Grade 2 | 38 | 28
  Pain: baseline Grade 3 | 6 | 17
  Pain: baseline Grade 4 | 7 | 3
  Pain: Total M12/ET | 413 | 417
  Pain: M12/ET None | 401 | 409
  Pain: M12/ET Grade 2 | 10 | 6
  Pain: M12/ET Grade 3 | 2 | 2
  Pain: M12/ET Grade 4 | 0 | 0

3. Secondary Outcome: Adult Mini-Rhinoconjuctivitis Quality of Life Questionnaire. Change From Baseline in RQLQ Score at Months 1,3,6,9 and 12/or Early Termination.
Description: The RQLQ consists of 7 domains rated on a 7-point scale with 0 being not troubled by the allergy symptoms,and 6 being extremely troubled. Total possible RQLQ score is 42 at any given evaluation. Scale of how troubled is:0=Not,2=Somewhat,3=Moderate,4=Quite a bit,5=Very,6 Extremely. Only change from baseline to month 12 primary analysis is provided.
Time Frame: baseline, months 1,3,6,9 and 12/or early termination
Population: Analysis is based on safety population, which is defined as subjects who took at least one dose of study medication.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Astepro Nasal Spray | Astelin Nasal Spray
Number analyzed (Participants) | 428 | 430
Units on a scale
  Baseline | 2.25 (1.103) | 2.18 (1.050)
  Month 1 | -0.77 (1.007) | -0.83 (0.959)
  Month 3 | -1.00 (1.063) | -1.00 (1.048)
  Month 6 | -1.04 (1.206) | -0.94 (1.230)
  Month 9 | -1.09 (1.228) | -1.16 (1.197)
  Month 12/Early termination | -0.88 (1.385) | -0.90 (1.339)
Statistical Analysis 1: Comparison: Astepro Nasal Spray vs Astelin Nasal Spray; Sample size was based on ICH Guideline E1:The Extent of Population Exposure to Assess Clinical Safety for Drugs Intended for Long-Term Treatment of Non-Life-Threatening Conditions. Comparisons performed using ANCOVA with baseline as a covariate. The model included treatment group and country as fixed effects to estimate least squares means; Test type: Superiority or Other; p = 0.368, ANOVA — This is the Baseline P-Value
Statistical Analysis 2: Comparison: Astepro Nasal Spray vs Astelin Nasal Spray; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.327, ANCOVA — This P-Value if for Month 1
Statistical Analysis 3: Comparison: Astepro Nasal Spray vs Astelin Nasal Spray; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.991, ANCOVA — This P-Value is for Month 3
Statistical Analysis 4: Comparison: Astepro Nasal Spray vs Astelin Nasal Spray; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.168, ANCOVA — This P-Value is for Month 6
Statistical Analysis 5: Comparison: Astepro Nasal Spray vs Astelin Nasal Spray; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.319, ANCOVA — This P-Value is for Month 9
Statistical Analysis 6: Comparison: Astepro Nasal Spray vs Astelin Nasal Spray; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.725, ANCOVA — This P-Value is for Month 12/ET

ADVERSE EVENTS:
Arm/Group | Astepro Nasal Spray | Astelin Nasal Spray
Serious Adverse Events (participants affected / at risk) | 7 | 10
Other Adverse Events (participants affected / at risk) | 163 | 146
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Astepro Nasal Spray | Astelin Nasal Spray
Battery change for internal cardiac defibrillator (Cardiac disorders) | 1/428 (1) | 0/430 (0)
Sialoadenitis (Infections and infestations) | 1/428 (1) | 0/430 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/428 (1) | 0/430 (0)
Acute Pyelonephritis (Infections and infestations) | 1/428 (1) | 0/430 (0)
Knee traumatism (Injury, poisoning and procedural complications) | 1/428 (1) | 0/430 (0)
Rectal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/428 (1) | 0/430 (0)
Exacerbation angina pectoris (Cardiac disorders) | 1/428 (1) | 0/430 (0)
Central Chest Pain (Cardiac disorders) | 1/428 (1) | 0/430 (0)
Exacerbation right shoulder pain (Musculoskeletal and connective tissue disorders) | 1/428 (1) | 0/430 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/428 (1) | 0/430 (0)
Removal of bladder stones (Renal and urinary disorders) | 0/428 (0) | 1/430 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 0/428 (0) | 1/430 (1)
Exertional dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/428 (0) | 1/430 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/428 (0) | 1/430 (1)
Pneumonia Chlamidalis (Infections and infestations) | 0/428 (0) | 1/430 (1)
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 0/428 (0) | 1/430 (1)
Fracture left foot (Injury, poisoning and procedural complications) | 0/428 (0) | 1/430 (1)
Broken nose (Injury, poisoning and procedural complications) | 0/428 (0) | 1/430 (1)
Syncope (Nervous system disorders) | 0/428 (0) | 1/430 (1)
Upper Abdominal Colic (Gastrointestinal disorders) | 0/428 (0) | 1/430 (1)
Total right hip replacement (Musculoskeletal and connective tissue disorders) | 0/428 (0) | 1/430 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Astepro Nasal Spray | Astelin Nasal Spray
Headache (Nervous system disorders) | 49/428 (49) | 43/430 (43)
Nasopharyngitis (Infections and infestations) | 34/428 (34) | 25/430 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29/428 (29) | 32/430 (32)
Dysgeusia (Nervous system disorders) | 28/428 (28) | 32/430 (32)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 23/428 (23) | 14/430 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies, joint publication is required to assure that the initial publication is based on all data from all sites and investigators participating in these studies agree not to present data gathered individually or by subgroup centers before the initial publication unless jointly agreed by all other investigators and the Sponsor. Authorship will be determined by mutual agreement.